CLINICAL TRIAL: NCT06122948
Title: Effect of Intranasal Midazolam Versus Ketamine Midazolam Combination as a Premedication in Children Undergoing Tonsillectomy and Adenoidectomy on the Occurrence of Postoperative Respiratory Adverse Events: a Double-blind, Randomized Controlled Trial
Brief Title: Effect of Intranasal Midazolam Versus Ketamine Midazolam Combination as a Premedication on the Occurrence of Postoperative Respiratory Adverse Events
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Khaled Abdelfattah Abdallah Sarhan, principal investigator, Asst. professor of anesthesia, Cairo university, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MD-227-2023
Record Dates: First submitted 2023-11-03; First posted 2023-11-08 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Tonsillectomy; Adenoidectomy; Drug-Related Side Effects and Adverse Reaction
Keywords: midazolam; ketamine; tonsillectomy; respiratory adverse events
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Intervention Model Description: Children will be randomly assigned to 2 groups: the midazolam group will receive intranasal midazolam (0.1 mg/kg), and the midazolam ketamine group will receive intranasal midazolam (0.1mg/kg) and ketamine (3mg/kg) for premedication
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The drug will be prepared by an anesthesia nurse who will not be involved in the study. The active drug will be administered by a fully trained anesthesiologist and Clear definitions of the respiratory adverse events will be provided to the involved anesthetist. All researchers directly involved in the study will be blinded to the drug which will be administered
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Group M) (Active Comparator): The midazolam group will receive intranasal midazolam (0.1 mg/kg)
  Interventions: Drug: The midazolam group
- (Group MK) (Experimental): Midazolam ketamine group will receive intranasal midazolam (0.1mg/kg) and ketamine (3mg/kg)
  Interventions: Drug: The midazolam ketamine group

INTERVENTIONS:
Drug: The midazolam group — The midazolam group will receive intranasal midazolam (0.1 mg/kg)
  Arms: (Group M)
Drug: The midazolam ketamine group — the midazolam ketamine group will receive intranasal midazolam (0.1mg/kg) and ketamine (3mg/kg)
  Arms: (Group MK)

SUMMARY:
The aim of this study is to investigate the effect of addition of intranasal ketamine to midazolam compared to midazolam alone as a premedication on the occurrence of PRAEs

DETAILED DESCRIPTION:
Perioperative respiratory adverse events (PRAEs) are the most common complication during pediatric anesthesia furthermore, most children presenting for AT have sleep-disordered breathing and obstructive sleep apnea syndrome (OSAS) caused by tonsillar hypertrophy which could aggravate the PRAEs specially with the use of the conventional sedatives as a premedication. A recent randomized controlled trial has shown that more than 50% of children premedicated with midazolam had experienced PRAEs . Midazolam and ketamine are commonly used as preoperative sedative drugs for pediatric populations. Ketamine is a safe and widely used sedative and analgesic in the pediatric emergency department (ED) with less profound effects on the upper airway and respiratory muscles. Intranasal ketamine administration is well tolerated and without serious adverse effects. The addition of ketamine to midazolam as a preoperative sedation to reduce the occurrence of PRAEs was not investigated before in children undergoing AT. The authors hypothesize that combination of ketamine to midazolam could offer optimum sedation condition while reducing the occurrence of PRAEs in children undergoing AT.

ELIGIBILITY:
Inclusion Criteria:

* Children both sexes male and female.
* Age from 3 to 12 years old.
* ASA grade I, II.
* undergoing elective AT procedures.

Exclusion Criteria:

* Congenital heart diseases (cyanotic and a cyanotic).
* Congenital syndromes affecting airway anatomy such as Pierre-Robin syndrome and Down syndrome.
* Severe lung diseases affecting either lung tissue such as pulmonary cystic fibrosis and idiopathic pulmonary fibrosis or affecting lung circulation such as pulmonary hypertension with marked limitation of Physical activity or inability to carry out any physical activity according to NHYA classification.
* Recent upper respiratory tract infection (less than two weeks).
* Neuromuscular diseases including cerebral palsy and epilepsy.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2023-11-04 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
The incidence of any perioperative respiratory adverse events (PRAEs) | 8 hours
  the incidence of any PRAEs (Perioperative respiratory adverse events (PRAEs) which are manifested as minor (oxygen desaturation (SaO2 less than 95% for 10 seconds) or coughing) and major as (bronchospasm, laryngospasm, airway obstruction, stridor or hypoxia (oxygen desaturation less than 90%)) among midazolam versus midazolam ketamine groups.

SECONDARY OUTCOMES:
Postoperative pain score | 8 hours
  • Postoperative pain score using (Wong-Baker Pain Scale)
Sedation success rate | 8 hours
  • Sedation success rate (score of 3 or 4 is considered successful sedation) using Funk score
Postoperative emergence delirium | 8 hours
  • Postoperative emergence delirium, a total Postoperative emergence delirium PAED score≥ 10 will be considered indicative of the presence of ED using (PAED scale

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university hospitals, kasralainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No